CLINICAL TRIAL: NCT02721186
Title: Effectiveness of Mass Drug Administration (MDA) for Reducing Seasonal Malaria Transmission Towards Its Elimination in Hotspot Areas in Zanzibar - a Cluster-randomised Controlled Trial
Brief Title: Effectiveness of Mass Drug Administration for Reducing Seasonal Malaria Transmission in Zanzibar
Acronym: MaDrAZ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ulrika Morris (Other)
Collaborators: Mahidol Oxford Tropical Medicine Research Unit (Other); RTI International (Other); The President's Malaria Initiative (Unknown); University of California, San Francisco (Other); Uppsala University (Other); Zanzibar Malaria Elimination Programme (Other Government)
Responsible Party: Sponsor-Investigator, Ulrika Morris, Postdoc, Study Coordinator, Karolinska Institutet
Organization: Karolinska Institutet (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MaDrAZ-001; ZAMREC/0001/January/2016 (Other: Zanzibar Medical Research Ethical Committee)
Record Dates: First submitted 2016-03-17; First posted 2016-03-29 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2017-10

CONDITIONS: Malaria; Plasmodium Infections
Keywords: Malaria; Plasmodium; Mass drug administration; Malaria elimination; Zanzibar; Dihydroartemisinin-Piperaquine; Single low dose Primaquine
MeSH Terms: conditions — Malaria | interventions — Mass Drug Administration; Single Person; Primaquine

ARMS (2):
- MDA with DHAp and SLD Primaquine (Experimental): MDA will be conducted at two time points with an approximate four-week interval. All consenting and eligible community members will be administered age-appropriate treatment dose of dihydroartemisinin-piperaquine (D-ARTEPP, Guilin Pharmaceutical (Shanghai) Co., Ltd., China) and single low dose (0.25mg/kg) primaquine (Primaquine, Remedica Ltd., Cyprus) in house-to-house campaigns.
  Interventions: Drug: MDA with DHAp and SLD Primaquine
- Control (No Intervention): The control arm (no MDA) will have the standard care offered by the Ministry of Health and Social welfare which applies to both arms. This includes passive case detection of individuals seeking treatment at local health facilities, and universal coverage of long lasting insecticide treated bed nets and indoor residual spraying in the study areas.

INTERVENTIONS:
Drug: MDA with DHAp and SLD Primaquine
  Other Names: Mass drug administration with DHAp and SLD Primaquine; MDA with Dihydroartemisinin-Piperaquine and SLD Primaquine; MDA with D-ARTEPP and single low dose Primaquine
  Arms: MDA with DHAp and SLD Primaquine

SUMMARY:
The overall aim of this study is to determine the effectiveness of two rounds of mass drug administration (MDA) with dihydroartemisinin-piperaquine (DHAp) + single low dose (SLD) primaquine for reducing seasonal malaria transmission in Shehias considered hotspots on Unguja Island, Zanzibar.

DETAILED DESCRIPTION:
Study design: This is a cluster-randomised controlled study with two arms: an intervention arm with two rounds of MDA with dihydroartemisinin-piperaquine (DHAp) + single low dose (SLD) primaquine, and a control arm with no MDA.

Study site and study population: The study will be conducted in 16 hotspot Shehias (8 Shehias randomly allocated to each arm), in three districts (West, Central and South districts) in Unguja Island, Zanzibar. Hotspot Shehias [Shehia being the smallest administrative structure in Zanzibar] are defined as Shehias with an annual malaria incidence of >0.8%, calculated as the number of confirmed malaria infections notified at health facilities and during active case detection in 2015 / Shehia projected population for 2015. The study population will include all consenting residents of the selected Shehias, reaching approximately 24000 people.

Study implementation: Two rounds of MDA with DHAp (D-ARTEPP, Guilin Pharmaceutical (Shanghai) Co., Ltd., China) and SLD (0.25mg/kg) primaquine (Primaquine, Remedica Ltd.,Cyprus ) will be conducted approximately four weeks apart in the intervention Shehias, at the anticipated lowest point of malaria transmission prior to the onset of malaria transmission associated with the main rains in April-June 2016. The first drug dose including DHAp and SLD primaquine will be given under supervision whenever possible; the other two doses of the standard once daily DHAp regimen will be taken unsupervised at home. Labelled packets containing all three doses will be left with the head of household with clear instructions for individuals not present at the time of the household visit.

Study objectives: The primary objective of the study is to determine the effectiveness of two rounds of MDA with DHAp + SLD primaquine for reducing seasonal malaria transmission in Shehias considered hotspots on Unguja Island, Zanzibar. The secondary objectives of the study include determining MDA coverage, compliance, and safety after one and two rounds of DHAp + SLD primaquine.

ELIGIBILITY:
Inclusion Criteria:

* Permanent or temporary resident of study Shehias (i.e., persons who stayed in the selected household the night before the interview)
* Provision of informed consent (refusal must be recorded)
* Age >6 months

Exclusion Criteria:

* Women pregnant in first trimester (assessed by a specific set of questions designed to exclude pregnancy)
* Severe disease that requires immediate referral to health facility or hospital
* Concurrent antimalarial treatment at time of MDA or during the last 14 days
* Inability to take oral medication

Additional exclusion criteria for treatment with SLD Primaquine:

* Pregnancy (all trimesters, assessed by a specific set of questions designed to exclude pregnancy)
* Women breast feeding infants aged < 6months

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 22500 (Actual)
Dates: Start 2016-04-30 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Cumulative notified malaria incidence in the MDA and control Shehias | 6 months after second round of MDA
  Cumulative notified malaria incidence determined as the number of confirmed malaria cases notified at health facilities (monitored through the malaria case notification system during the period of six months) over the Shehia population size determined by population enumeration at the time of the intervention.

SECONDARY OUTCOMES:
PCR determined community prevalence of Plasmodium infections in the MDA and control Shehias | Baseline and 3 months after second round of MDA
  PCR determined community prevalence of Plasmodium infections determined by cross-sectional screening in every other household in the study area at the time of the first round of MDA, and at six months after the second round of MDA.

OTHER OUTCOMES:
Population coverage of the MDA intervention at each round | Through completion of first and second round of MDA, i.e. 15 days and 48 days after initiation of MDA, respectively.
  MDA coverage determined as the number of administered DHAp and SLD primaquine doses during the first and second round of MDA, over over the Shehia population size determined by population enumeration at the time of the intervention.
Proportion of population receiving two rounds of MDA | Through completion of the second round of MDA, i.e. 48 days after initiation of MDA.
  The proportion of the population having received zero, one or two rounds of MDA. Refusal and reason for refusal to participate will be recorded.
Population compliance to the MDA intervention at each round | 7 days after both first and second round of MDA
  MDA compliance, i.e. the proportion of the population that have taken one, two or all three doses of DHAp + SLD primaquine, will be evaluated in a subset of the population by post-MDA surveys conducted seven days after the initiation of each MDA round. The post MDA surveys will include both a questionnaire and finger prick blood sampling for measuring piperaquine blood concentrations.
Occurence of adverse events after MDA with DHAp and SLD primaquine | 14 days after both first and second round of MDA
  A brief questionnaire will be conducted in a subset of the population during post-MDA surveys conducted seven days after the initiation of each MDA round. The questionnaire will include specific questions regarding adverse events such as vomiting, nausea, gastrointestinal upset, rash and fatigue. Severe adverse events, especially symptoms of haemolysis, will be captured at health facilities where haemoglobin and dark urine (representing haemolysis) will be measured and reported using the pharmacovigilance forms and the Primaquine Roll Out Monitoring Pharmacovigilance Tool (PROMPT) developed by the Global Health Group at University of California San Francisco.
Cumulative notified malaria incidence in the MDA and control Shehias during the following high transmission season. | 15 months after second round of MDA
  Cumulative notified malaria incidence during the following high transmission season, monitored through the malaria case notification system, to assess the long-term effectivness of MDA.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Björkman, MD, PhD, Principal Investigator — Karolinska Institutet; Abdullah S Ali, Programme Manager, Principal Investigator — Zanzibar Malaria Elimination Programme
Locations (1):
- Zanzibar Malaria Elimination Programme, Mwanakwerekwe, Urban District, Zanzibar, Tanzania

REFERENCES:
- [Derived] Shah MP, Hwang J, Choi L, Lindblade KA, Kachur SP, Desai M. Mass drug administration for malaria. Cochrane Database Syst Rev. 2021 Sep 29;9(9):CD008846. doi: 10.1002/14651858.CD008846.pub3. PMID 34585740
- [Derived] Morris U, Msellem MI, Mkali H, Islam A, Aydin-Schmidt B, Jovel I, Shija SJ, Khamis M, Ali SM, Hodzic L, Magnusson E, Poirot E, Bennett A, Sachs MC, Tarning J, Martensson A, Ali AS, Bjorkman A. A cluster randomised controlled trial of two rounds of mass drug administration in Zanzibar, a malaria pre-elimination setting-high coverage and safety, but no significant impact on transmission. BMC Med. 2018 Dec 10;16(1):215. doi: 10.1186/s12916-018-1202-8. PMID 30526588